CLINICAL TRIAL: NCT00679276
Title: Treatment Outcomes of Vaginal Prolapse Repair
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Predeep Nagaraju, MD, William Beaumont Hospital
Other Study IDs: 2008-102
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-06

CONDITIONS: Vaginal Prolapse
Keywords: vaginal prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients having surgical repair of a vaginal prolapse .
  Interventions: Procedure: Prolift

INTERVENTIONS:
Procedure: Prolift — surgical repair of vaginal prolapse

SUMMARY:
Chart review conducted on all patients having had Prolift surgery since 2005 by Dr. Lary Sirls, Dr. Predeep Nagaraju and Dr. Kenneth Peters at William Beaumont Hospital.

DETAILED DESCRIPTION:
Chart review conducted on all patients having had Prolift surgery since 2005 by Dr. Lary Sirls, Dr. Predeep Nagaraju and Dr. Kenneth Peters at William Beaumont Hospital. Preoperative, intraoperative and post-operative data will be collected from the hospital and physician medical records. A questionnaire will be mailed to patients whose charts have been reviewed to assess urinary and bowel function, satisfaction with treatment and changes in sexual function. Completion of the questionnaire is voluntary.

ELIGIBILITY:
Inclusion Criteria:

* Women having Prolift repair at William Beaumont Hospital

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having prolift surgery at William Beaumont Hospital by Dr. Lary Sirls, Dr. Predeep Nagaraju, and Dr. Kenneth Peters.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Predeep Nagaraju, MD, Principal Investigator — Corewell Health East